CLINICAL TRIAL: NCT06972238
Title: A Prospective Observational Study of Acute Pancreatitis Severity and the Association of Glucose Time in Range and Stress Hyperglycaemia, Plasma Insulin Depletion and Bacterial Endotoxaemia
Brief Title: Glucose Levels in Acute Pancreatitis and the Impact of Insulin Depletion and Bacterial Endotoxaemia
Acronym: GLIDE
Status: Not yet recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B02533; B02533 (Other: Manchester University NHS Foundation Trust)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pancreatitis, Acute; Hyperglycaemia
Keywords: Pancreatitis; Hyperglycaemia; inflammation; clinical severity; beta-cell
MeSH Terms: conditions — Pancreatitis; Hyperglycemia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are currently no early predictive biomarkers for severity of acute pancreatitis (AP) that would allow stratification of patients for potential early interventional therapies. Hyperglycaemia is frequently observed to accompany and contribute to severe AP. However, the underlying mechanism is multifactorial, including in the acute phase of injury, where elevated adrenaline, cortisol and glucagon and inflammatory cytokine-induced insulin resistance all contribute to hyperglycaemia. The investigators propose that the extent of collateral injury of pancreatic β-cells and consequent loss of insulin secretion during the course of acute pancreatitis (AP) underlies disease severity. The investigators will measure plasma C-peptide (as a reliable readout of endogenous insulin), with moment-to-moment glucose monitoring (using subcutaneous continuous glucose monitoring devices), and bacterial endotoxin (lipopolysaccharide (LPS) in a prospective cohort of 30 severe AP patient blood samples taken every 5 days for up to 5 weeks of hospitalization.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is associated with metabolic dysregulation including dysglycaemia which may predict poor clinical outcomes. Continuous glucose monitoring (CGM) offers a novel method for assessing glycaemia continuously in real time. The percentage of time spent in normal glucose range (TIR; 3.9-10.0 mmol/L) may correlate with key outcomes, including length of hospital stay (LOS), need for critical care, and mortality. This study aims to evaluate whether TIR measured via CGM can serve as a predictive marker in AP management.

While hyperglycaemia is frequently observed to accompany and contribute to severe AP, the underlying mechanism is not fully understood and is likely to be multifactorial and change over the disease course. For example, in the acute phase of injury, the elevated adrenaline, cortisol and glucagon and inflammatory cytokine-induced insulin resistance contribute to hyperglycaemia. The investigators propose that later in the course, the extent of collateral injury of pancreatic β-cells and consequent loss of insulin secretion may also impact disease severity. This loss of insulin secretion leads to the loss of insulin-mediated pancreatic antimicrobial secretion into the gut leading to gut dysbiosis, inflammation, reduced barrier function, bacterial translocation and infected pancreatic necrosis, resulting in severe AP. This suggests that plasma insulin depletion (with extensive hyperglycaemia) may represent early predictive biomarkers and elevated plasma bacterial endotoxin may represent a late biomarker for disease severity.

This is a single-centre, single-arm, non-randomised, observational study of adults (18 years and older) admitted to Manchester Royal Infirmary with acute pancreatitis. The study aims to recruit 30 participants over 12 months. The study's primary objective is to determine the overall time spent in normal glucose range (TIR; 3.9-10.0 mmol/L) in patients admitted with acute pancreatitis. Secondary objectives include:

1. Evaluating the association between TIR and clinical severity of acute pancreatitis.
2. Evaluating the association between TIR and length of hospital stay.
3. Determining the relationship between changes in plasma c-peptide and bacterial endotoxin with clinical severity of acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or over
2. Admission diagnosis of acute pancreatitis (based on Revised Atlanta Criteria)
3. Ability to provide informed consent in English

Exclusion Criteria:

1. Known diabetes mellitus
2. Use of insulin therapy before admission
3. Pregnancy
4. Contraindications to CGM (e.g., allergy to device adhesive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on the surgical and medical wards at Manchester Royal Infirmary, (Manchester University NHS Foundation Trust [MFT]). Adults with acute pancreatitis will be recruited following admission to hospital under the treating clinical team. Patients will be identified by a member of the usual clinical team based upon analysis of the acute surgical take on our electronic health record (HIVE), cross referencing abdominal pain and raised lipase and imaging when appropriate.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Time in range | 28 days
  The primary outcome is time spent in normal range (3.9 - 10.0 mmol/l) based on CGM sensor glucose levels during inpatient stay

SECONDARY OUTCOMES:
Endogenous beta-cell insulin secretion | 28 days
  Plasma c-peptide
Bacterial endotoxin levels | 28 days
  Plasma bacteria endotoxin
Clinical severity of acute pancreatitis | 28 days
  BISAP Score

CONTACTS AND LOCATIONS:
Overall Officials: Hood M Thabit, Principal Investigator — Manchester Royal Infirmary

IPD SHARING:
Plan to Share IPD: Yes
Anonymised primary and secondary endpoints data, following reasonable request.
Supporting Information: CSR
Time Frame: 12 months following study completion.
Access Criteria: Following reasonable request to the researcher by email.